CLINICAL TRIAL: NCT00323154
Title: Nalbuphine for the Treatment of Opioid Induced Pruritus in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Carolyne Montgomery, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C02-0589; W02-0175
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Pruritis
Keywords: Morphine, analgesia
MeSH Terms: conditions — Pruritus; Agnosia | interventions — Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Nalbuphine

SUMMARY:
Itching is a frequent and disturbing side effect of the use of pain medication such as morphine. In the post-operative period, it can be more distressing to pediatric patients than their pain. The current first line treatment, an antihistamine (Benadryl), has a low efficacy. This treatment causes sleepiness and may be dangerous when used in combination with other drugs.

Nalbuphine has analgesic properties similar to morphine as well as the ability to reverse some morphine-induced side effects, such as respiratory depression and itching. Nalbuphine has been used effectively for patients undergoing Caesarean sections. However, the effectiveness of nalbuphine in the pediatric population has not been investigated.

We want to determine the efficacy of nalbuphine in the treatment of itching after morphine for postoperative pain relief. We will use a novel method to measure the effect of the treatment using an intensity scale before and after the drug, to determine the intensity difference.

DETAILED DESCRIPTION:
PURPOSE Primary To determine the efficacy of nalbuphine (50 - 100 mcg/kg intravenously) in the treatment of opioid induced pruritus in a multi-center tertiary care pediatric patient population.

Secondary Determine the effect of treatment with nalbuphine on a subjects analgesia and level of sedation.

HYPOTHESIS

Primary Outcome:

Nalbuphine will be effective in the treatment of opioid induced pruritus; a 50% reduction in pruritus intensity will be considered clinically significant.

Secondary Outcome:

Treatment with nalbuphine will not result in attenuation of analgesia or an increase in sedation

JUSTIFICATION Itch is a frequent and disturbing side effect of opioid use. A recent internal review of the pediatric pain service at the University of Alberta Hospital, Edmonton, Alberta found a 40% incidence of pruritus in patients receiving opioids. A similar review at British Columbia Children's Hospital demonstrated a 22% of patients incidence of pruritus.

OBJECTIVES The compare the efficacy of nalbuphine to placebo for the treatment of opioid-induced pruritus. It is anticipated that nalbuphine will result in a greater than 50% reduction in pruritus intensity.

RESEARCH METHOD This study will be a randomized, double-blinded, placebo controlled trial of nalbuphine for the treatment of opioid-induced pruritus. Pruritus intensity will be measured using a standardized assessment tool / Color Analog Scale (CAS). This is a metric scale which will be used to quantify pruritus on a scale of zero to ten. Using this scale a score of zero is represented by white, increasing pruritus severity being represented by darker shades of the color red, along a ruler.

Data analysis will be based on intenton to treat. It will be a multi-center study involving tertiary care centers with acute pediatric pain services.

Subjects will be divided into two groups by computer generated block randomization; one group will receive treatment with nalbuphine while the other will receive placebo. The patient and investigator will be blinded to the treatment administered.

REASON FOR PLACEBO CONTROLLED STUDY DESIGN Current first line therapy for opioid induced pruritus, with diphenhydramine is associated with a low efficacy (33%) (1). Recognizing that there can be up to 30% self report response to placebo, it is felt that conducting this study as a placebo-controlled trial will be necessary for the demonstration of significant improvement in pruritus intensity.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative morphine administration

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Estimated)
Dates: Start 2004-03; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Pruritis intensity

SECONDARY OUTCOMES:
Pain, sedation

CONTACTS AND LOCATIONS:
Overall Officials: Carolyne Montgomery, MD, Principal Investigator — The University of British Columbia
Locations (1):
- British Columbia's Children's Hospital, Vancouver, British Columbia, Canada